CLINICAL TRIAL: NCT02072239
Title: First-In-Human Study to Demonstrate the Preliminary Safety and Efficacy of the Angioshield System to Provide Mechanical Support for Vein Grafts Used in CABG Surgery
Brief Title: Angioshield First-In-Human Study to Demonstrate the Preliminary Safety and Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neograft Technologies, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP11-002
Record Dates: First submitted 2014-02-13; First posted 2014-02-26 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Intimal Hyperplasia; Atherosclerosis; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device Applied (Experimental): All participants will be treated with the Angioshield
  Interventions: Device: Angioshield

INTERVENTIONS:
Device: Angioshield — The Angioshield wrap provides external structural support for the saphenous vein graft used in CABG surgery and is intended to prevent over distention of the graft under arterial pressure, potentially improving graft patency and reducing the likelihood of graft failure.

SUMMARY:
The purpose of this study is to determine whether or not the Angioshield device can be safely applied to support saphenous vein grafts used in standard coronary bypass surgery.

DETAILED DESCRIPTION:
\This is a first in human study which is intended to determine if a larger pivotal study is justified.

ELIGIBILITY:
Inclusion Criteria:

Subject will be eligible for inclusion in the investigation if he/she:

* is between the ages of 18 and 80 years of age, inclusive
* requires Coronary Atery Bypass Graft (CABG) surgery with minimum of one SVG used to bypass a stenosis in the Right Coronary, the Circumflex, a Diagonal, or an Obtuse Marginal artery, due to atherosclerotic coronary artery disease
* is able to give their informed written consent
* is willing and able to complete all follow-up visits and procedures

Exclusion Criteria:

Subject will be excluded from participation in the investigation if he/she:

* is currently enrolled in another clinical investigation
* is unable to tolerate or comply with required post-surgical medications or imaging (e.g., anticoagulation regimen; or known allergy to contrast agent)
* is or may be pregnant or is lactating, or plans to become pregnant in the next 12 months
* shows a presence of hypercoagulable state or history of idiopathic venous or arterial thrombosis
* has had an acute MI within the last 21 days
* has had a previous CABG
* requires emergency surgery
* has a left ejection fraction (LEF) less than 20%
* has a target vessel stenosis of less than 70%
* has a transmural infarct of the target artery territory
* currently requiring dialysis
* is having concomitant-surgery of any kind
* has varicose veins
* has had previous saphenectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days
  The primary objective of this study is to provide acute and subacute (up to 30 days) safety outcomes to support expansion to a pivotal study involving a larger subject population. All Major Adverse Cardiac Events (MACE), defined as the composite of cardiac death, myocardial infarction (Q-wave and non-Q wave), and target vessel revascularization, will be evaluated at 30 days post-operative.

SECONDARY OUTCOMES:
MACE and Graft Patency | 30, 90 and 365 Days
  The secondary objective of this study is to assess long term (up to 1 year) safety outcomes and vein patency for additional safety and preliminary efficacy information. All MACE, defined as the composite of cardiac death, myocardial infarction (Q-wave and non-Q wave), and target vessel revascularization will be evaluated at 90 and 365 days and to assess patency of the treated saphenous vein graft at 30, 90 and 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sadowski, MD, PhD, Principal Investigator — Pope John Paul II Hospital and Cardiology Collegium Medicum Jagiellonian University, Krakow, Poland
Locations (1):
- Pope John Paul II Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No